CLINICAL TRIAL: NCT00001696
Title: A Pharmacokinetic Study of Genistein, a Tyrosine Kinase Inhibitor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980099; 98-C-0099
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-04

CONDITIONS: Cancer
Keywords: Anti-metastatic; Chemoprevention; Isoflavinoid; Prostate Cancer; Signal Transduction
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — Genistein

INTERVENTIONS:
Drug: Genistein

SUMMARY:
Genistein is a natural product found in soy beans; its consumption has been associated with a low incidence of metastatic prostate cancer. Genistein is a known protein-tyrosine kinase inhibitor, and in preclinical studies it has been shown to increase cell adhesion. Increases in cell adhesion in vivo would phenotypically reverse the first step in the metastatic cascade, potentially preventing metastasis formation, and is consistent with epidemiologic findings. This study seeks to determine the pharmacokinetics of genistein in humans by administering a single dose of genistein and performing a pharmacokinetic analysis. Patients will be treated with two formulations of genistein (a 43% genistein preparation or a 90% preparation). This is a phase I study, and patients will be treated on one of three dosing levels. Patients will be randomly assigned to receive one formulation first, followed by a washout period, and will then receive the second preparation (i.e. a randomized cross over design). Information from this study will be used to optimally design a multiple dose study wherein patients will be treated for longer periods of time.

DETAILED DESCRIPTION:
Genistein is a natural product found in soy beans; its consumption has been associated with a low incidence of metastatic prostate cancer. Genistein is a known protein-tyrosine kinase inhibitor, and in preclinical studies it has been shown to increase cell adhesion. Increases in cell adhesion in vivo would phenotypically reverse the first step in the metastatic cascade, potentially preventing metastasis formation, and is consistent with epidemiologic findings. This study seeks to determine the pharmacokinetics of genistein in humans by administering a single dose of genistein and performing a pharmacokinetic analysis. Patients will be treated with two formulations of genistein (a 43% genistein preparation or a 90% preparation). This is a phase I study, and patients will be treated on one of three dosing levels. Patients will be randomly assigned to receive one formulation first, followed by a washout period, and will then receive the second preparation (i.e., a randomized cross over design). Information from this study will be used to optimally design a multiple dose study wherein patients will be treated for longer periods of time. The duration of this study is estimated to be about 4 weeks long for each patient.

ELIGIBILITY:
Must be 18 years old or greater.

ECOG performance status of 0-1.

Individuals without a history of cancer are eligible, as are those with a history of cancer. Individuals with a history of cancer (excluding non-melanomatous skin cancer ) will need to submit their pathology slides for review in the Laboratory of Pathology, NCI.

Must be able to understand and give informed consent.

Life expectancy greater than 6 months.

Hgb greater than or equal to 8.0gm/dl, platelets greater than or equal to 100,000/microliters, ANC greater than or equal to 1000/microliters, creatinine less than or equal to 2.0/mg/dl, SGPT and SGOT less than or equal to 147 and 168 U/L, total bilirubin less than or equal to 2 mg/dl (patients with a higher level of bilirubin due to a familial defect in bilirubin metabolism will be considered on an individual basis).

No history of breast cancer.

No pregnant or breast feeding subjects.

Must not be HIV positive.

No history of venous thrombosis within the past year.

No medical conditions, which, in the opinion of the investigators would jeopardize either the patient or the integrity of the data obtained.

No patients who are currently receiving active therapy for neoplastic disorders. However, patients with prostate cancer who are on an LHRH agonist (e.g., Lupron or Zoladex), or who have undergone surgical castration, are eligible for study.

No patients who are on estrogen therapy.

No patients taking hormonal forms of contraception.

No patients with a known soy intolerance.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15
Dates: Start 1998-04; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Severson RK, Nomura AM, Grove JS, Stemmermann GN. A prospective study of demographics, diet, and prostate cancer among men of Japanese ancestry in Hawaii. Cancer Res. 1989 Apr 1;49(7):1857-60. PMID 2924323
- [Background] Adlercreutz H. Western diet and Western diseases: some hormonal and biochemical mechanisms and associations. Scand J Clin Lab Invest Suppl. 1990;201:3-23. PMID 2173856
- [Background] Adlercreutz H, Markkanen H, Watanabe S. Plasma concentrations of phyto-oestrogens in Japanese men. Lancet. 1993 Nov 13;342(8881):1209-10. doi: 10.1016/0140-6736(93)92188-y. PMID 7901532